CLINICAL TRIAL: NCT04077840
Title: Autoimmune Diseases and Serum Autoantibodies in Non-celiac Wheat Sensitivity Patients in Comparison to IBS Patients
Brief Title: Autoimmune Diseases and Serum Autoantibodies in NCWS and IBS Patients
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Clinical Professor, University of Palermo
Other Study IDs: ACPM22
Record Dates: First submitted 2019-08-31; First posted 2019-09-04 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Non-celiac Gluten Sensitivity; Non-celiac Wheat Sensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NCGS/NCWS patients: Adult patients with a definitive diagnosis of NCWS, based on DBPC wheat challenge, most of them suffering from IBS-like-clinical presentation, according to Rome IV criteria. The patients were consecutively recruited between January 2016 and October 2017 at the outpatient clinics of the Department of Internal Medicine of the University Hospital of Palermo and the Department of Internal Medicine of the Hospital of Sciacca (both in southern Italy)
- Heathy blood donors: Consecutive healthy blood donors sex- (+ 5%) and age-matched (+ 2 years) with the NCWS patients.
- IBS patients: Consecutive patients with a diagnosis of IBS unrelated to NCWS or other types of food "intolerance/allergy", who were consecutively recruited during the study period and sex- (+ 5%) and age-matched (+ 2 years) with the NCWS patients.

SUMMARY:
In recent years, a new gluten- or wheat-related disease has emerged, a condition labelled "non-celiac gluten sensitivity" (NCGS) or "non-celiac wheat sensitivity" (NCWS). Given the lack of a diagnostic biomarker, NCGS/NCWS mostly remains a diagnosis of exclusion, especially respect to CD and WA, so a confirmatory test is required. The Salerno experts suggested the double-blind, placebo-controlled (DBPC), cross-over, gluten/wheat challenge as the gold standard test to discriminate true NCGS/NCWS patients. There are conflicting data about the real mechanisms which induce symptoms in NCGS/NCWS patients after wheat ingestion. Some Authors suggested a prevalent role for Fermentable Oligosaccharides-Disaccharides-Monosaccharides and Polyols (FODMAPs), rather than gluten in determining the symptoms. Other studies underlined the activation of mechanisms of both innate and acquired immunity in NCWS patients, after wheat ingestion. In the present study, we included a group of consecutive NCWS patients, diagnosed with DBPC wheat challenge, to evaluate a) the frequency of autoimmune diseases, b) the frequency and pattern of serum ANA and other non-organ-specific and/or organ-specific autoantibodies, and c) the possible correlations between autoimmune diseases and serum autoantibodies presence and other NCWS-related disease characteristics, in comparison with age- and sex- matched healthy blood donors and IBS patients unrelated to NCWS.

DETAILED DESCRIPTION:
In recent years, a new gluten- or wheat-related disease has emerged, a condition labelled "non-celiac gluten sensitivity" (NCGS) or "non-celiac wheat sensitivity" (NCWS). This is very often a self-reported condition, since patients refer to intestinal (mainly irritable bowel syndrome (IBS)-like) and/or extra-intestinal symptoms (i.e. fatigue, headache) caused by gluten or wheat ingestion, even though they do not have celiac disease (CD) or wheat allergy (WA). Given the lack of a diagnostic biomarker, NCGS/NCWS mostly remains a diagnosis of exclusion, especially respect to CD and WA, so a confirmatory test is required. The Salerno experts suggested the double-blind, placebo-controlled (DBPC), cross-over, gluten/wheat challenge as the gold standard test to discriminate true NCGS/NCWS patients.

However, there are conflicting data about the real mechanisms which induce symptoms in NCGS/NCWS patients after wheat ingestion. Some Authors suggested a prevalent role for Fermentable Oligosaccharides-Disaccharides-Monosaccharides and Polyols (FODMAPs), rather than gluten in determining the symptoms. Other studies underlined the activation of mechanisms of both innate and acquired immunity in NCWS patients, after wheat ingestion. In line with the evidence of an immunologic activation in NCWS, we showed in a previous study that about one quarter of NCWS patients suffered from associated autoimmune diseases (mainly Hashimoto's thyroiditis), compared with a smaller proportion of a control group including IBS patients (about 3%). Furthermore, we showed that serum samples of NCWS patients tested positive for anti-nuclear (ANA) in more than one third of the cases. However, that study included mainly patients evaluated in a retrospective manner and no other autoantibodies were evaluated apart from ANA.

In the present study, we included a group of consecutive NCWS patients, diagnosed with DBPC wheat challenge, to evaluate a) the frequency of autoimmune diseases, b) the frequency and pattern of serum ANA and other non-organ-specific and/or organ-specific autoantibodies, and c) the possible correlations between autoimmune diseases and serum autoantibodies presence and other NCWS-related disease characteristics, in comparison with age- and sex- matched healthy blood donors and IBS patients unrelated to NCWS.

ELIGIBILITY:
NCWS

Inclusion criteria:

* resolution of symptoms on a standard elimination diet, without wheat, cow's milk, yeast, and other food(s) causing self-reported symptoms
* symptom reappearance on a DBPC wheat challenge. As in previous studies, a DBPC cow's milk protein challenge and other open food challenges were also performed
* age above 18 years and <65 years
* follow-up duration longer than 12 months after the initial diagnosis
* at least two outpatient visits during the follow-up period.

Exclusion criteria:

* positive serum assays for celiac disease (i.e. anti-tissue transglutaminase (anti-tTG) IgA and anti-deamidated gliadin peptides (anti-DGP) IgG antibodies)
* presence of intestinal villous atrophy, documented in all the patients carrying the DQ2 and/or the DQ8 HLA haplotypes
* positive IgE-mediated immune-allergy tests to wheat (skin prick tests and/or specific serum IgE detection).

IBS IBS diagnosis had been made in accordance with the Rome IV criteria and none of these patients improved on an elimination diet without wheat, cow's milk, egg, tomato or chocolate.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We prospectively surveyed 58 adult patients with a definitive diagnosis of NCWS, based on DBPC wheat challenge, most of them suffering from IBS-like-clinical presentation, according to Rome IV criteria. The patients were consecutively recruited between January 2016 and October 2017 at the outpatient clinics of the Department of Internal Medicine of the University Hospital of Palermo and the Department of Internal Medicine of the Hospital of Sciacca (both in southern Italy). Two control groups were selected. One included 76 consecutive healthy blood donors sex- (+ 5%) and age-matched (+ 2 years) with the NCWS patients, while the second included 55 patients with a diagnosis of IBS unrelated to NCWS or other types of food "intolerance/allergy", who were consecutively recruited during the study period and sex- (+ 5%) and age-matched (+ 2 years) with the NCWS patients.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Frequency of associated autoimmune diseases | 22 months
  The presence of autoimmune disorders both in NCWS and IBS control patients was evaluated by a structured questionnaire and a review of patients' clinical records. The presence of one of the following was looked for in all subjects: connective tissue diseases, autoimmune endocrinological diseases, autoimmune hepatitis, primary biliary cirrhosis, epilepsy with cerebral calcification, unexplained cerebellar ataxia, alopecia, psoriasis, atrophic autoimmune gastritis, and immune anemia, neutropenia, or thrombocytopenia.
Serum autoantibodies | 22 months
  The frequency, titers and patterns of serum ANA, antibodies against double stranded DNA (anti-dsDNA), extractable nuclear antigen (ENA), islet cells of the pancreas (ICA), parietal cell antibodies (APCA), and, finally, tireoglobulin (anti-TG) and thyroid peroxidase (anti-TPO) were evaluated by ELISA and Immunofluorescence.
Clinical characteristics of NCWS and IBS patients | 22 months
  Frequency of autoimmune diseases and autoantibodies were correlated with the following clinical and laboratory parameters: age at diagnosis, gender, coexistent pathologies, atopic diseases and nickel allergy, anemia, coexistent other food allergies, presence of IBS-like symptoms, functional dyspepsia, and extraintestinal symptoms, BMI, duodenal histology lesions, and DQ2/DQ8 HLA haplotypes.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Department of Internal Medicine, University Hospital of Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carroccio A, D'Alcamo A, Cavataio F, Soresi M, Seidita A, Sciume C, Geraci G, Iacono G, Mansueto P. High Proportions of People With Nonceliac Wheat Sensitivity Have Autoimmune Disease or Antinuclear Antibodies. Gastroenterology. 2015 Sep;149(3):596-603.e1. doi: 10.1053/j.gastro.2015.05.040. Epub 2015 May 27. PMID 26026392
- [Result] Carroccio A, Mansueto P, D'Alcamo A, Iacono G. Non-celiac wheat sensitivity as an allergic condition: personal experience and narrative review. Am J Gastroenterol. 2013 Dec;108(12):1845-52; quiz 1853. doi: 10.1038/ajg.2013.353. Epub 2013 Nov 5. PMID 24169272
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Catassi C, Elli L, Bonaz B, Bouma G, Carroccio A, Castillejo G, Cellier C, Cristofori F, de Magistris L, Dolinsek J, Dieterich W, Francavilla R, Hadjivassiliou M, Holtmeier W, Korner U, Leffler DA, Lundin KE, Mazzarella G, Mulder CJ, Pellegrini N, Rostami K, Sanders D, Skodje GI, Schuppan D, Ullrich R, Volta U, Williams M, Zevallos VF, Zopf Y, Fasano A. Diagnosis of Non-Celiac Gluten Sensitivity (NCGS): The Salerno Experts' Criteria. Nutrients. 2015 Jun 18;7(6):4966-77. doi: 10.3390/nu7064966. PMID 26096570
- [Result] Di Liberto D, Mansueto P, D'Alcamo A, Lo Pizzo M, Lo Presti E, Geraci G, Fayer F, Guggino G, Iacono G, Dieli F, Carroccio A. Predominance of Type 1 Innate Lymphoid Cells in the Rectal Mucosa of Patients With Non-Celiac Wheat Sensitivity: Reversal After a Wheat-Free Diet. Clin Transl Gastroenterol. 2016 Jul 7;7(7):e178. doi: 10.1038/ctg.2016.35. PMID 27388423
- [Result] Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology. 2016 Feb 19:S0016-5085(16)00223-7. doi: 10.1053/j.gastro.2016.02.032. Online ahead of print. PMID 27144617
- [Result] Losurdo G, Principi M, Iannone A, Giangaspero A, Piscitelli D, Ierardi E, Di Leo A, Barone M. Predictivity of Autoimmune Stigmata for Gluten Sensitivity in Subjects with Microscopic Enteritis: A Retrospective Study. Nutrients. 2018 Dec 18;10(12):2001. doi: 10.3390/nu10122001. PMID 30567296
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Sapone A, Bai JC, Ciacci C, Dolinsek J, Green PH, Hadjivassiliou M, Kaukinen K, Rostami K, Sanders DS, Schumann M, Ullrich R, Villalta D, Volta U, Catassi C, Fasano A. Spectrum of gluten-related disorders: consensus on new nomenclature and classification. BMC Med. 2012 Feb 7;10:13. doi: 10.1186/1741-7015-10-13. PMID 22313950